CLINICAL TRIAL: NCT07046585
Title: Evaluation of the Natera Colorectal Cancer Screening Test in an Average Risk Population (FIND-CRC)
Acronym: FIND-CRC
Status: Recruiting | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 25-080-ECP
Record Dates: First submitted 2025-06-13; First posted 2025-07-01 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Colo-rectal Cancer
Keywords: colorectal cancer; colon cancer; early cancer detection
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants at average risk for colorectal cancer: Participants 40 years of age or older at time of consent, planning or intending to undergo asymptomatic screening colonoscopy.

SUMMARY:
The FIND-CRC study is a prospective collection of samples and data from participants who are at average risk of developing colorectal cancer (CRC). Collected samples and data will be analyzed to evaluate the clinical performance of the Natera CRC Screening Test.

DETAILED DESCRIPTION:
Participants who meet study inclusion criteria will be invited to enroll in the study and will provide written consent prior to study procedures. Participants will provide blood samples and will be required to have a colonoscopy performed within 120 days of their blood draw. No test results from the blood collection will be provided to participants or clinicians.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. 40 years of age or older at the time of consent.
3. Planning or intending to undergo a standard of care colonoscopy.
4. Able to tolerate venipuncture for research draw(s).
5. Able and willing to provide blood samples within the 120 days prior to a standard-of-care pre-bowel preparation procedure and colonoscopy procedure.
6. Willing and able to comply with the study visit schedule and study requirements.

Exclusion Criteria:

1. Any prior history of any kind of malignancy (exception: participants who have undergone surgical removal of skin squamous cell or basal cell cancers may be enrolled, provided the procedure was completed at least 12 months prior to consent for the study).
2. Had a complete colonoscopy with adequate bowel preparation in the previous nine (9) years.
3. Undergoing diagnostic colonoscopy for the investigation of symptoms.
4. Up to date with colorectal cancer screening from any non-invasive test.
5. Precancerous findings on most recent colonoscopy.
6. Had a prior colorectal resection for any reason other than sigmoid diverticular disease.
7. Known personal history of any of the following high-risk conditions:

7a. Inflammatory bowel disease. 7b. Known hereditary condition that would increase risk of colorectal cancer (example Lynch Syndrome).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants 40 years of age or older who are at average risk of colorectal cancer and scheduled for a screening colonoscopy as part of their standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-07-10 (Estimated); Study Completion 2033-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 24 months
  The primary outcomes of this study are sensitivity of the Natera CRC Screening Test for the detection of colorectal cancer (CRC) and specificity of the test for advanced neoplasia (AN), as assessed by agreement of the Natera CRC Screening test with colonoscopy findings.

SECONDARY OUTCOMES:
Secondary Outcomes | 24 months
  The secondary outcomes of this study are sensitivity and specificity of the Natera CRC Screening Test for the detection of Advanced Precancerous Lesions (APL) and specificity of the test for Negative findings, as assessed by agreement of the Natera CRC Screening test with colonoscopy findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Natera, Inc, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No